CLINICAL TRIAL: NCT05716087
Title: An Open Label, Single Arm, Multicenter Phase II Study of the Efficacy and Safety of Rocbrutinib Monotherapy for Recurrent or Refractory Mantle Cell Lymphoma
Brief Title: A Study of Rocbrutinib in Participants With Relapse or Refractory Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Lupeng Pharmaceutical Company LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP-168-CN201
Record Dates: First submitted 2023-01-19; First posted 2023-02-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Mantle Cell Lymphoma (MCL)
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rocbrutinib (Experimental): Subjects who have previously received BTK inhibitors treatment failed or relapsed after remission or intolerated
  Interventions: Drug: Rocbrutinib

INTERVENTIONS:
Drug: Rocbrutinib — Subjects to take Rocbrutinib tablets orally with 240mL water, without food, Once daily.The treatment will continue until progressive disease, unacceptable toxicity, etc.
  Other Names: NWP-775; LP-168

SUMMARY:
This is an open-label, single arm, multi-center Phase 2 study of oral Rocbrutinib in patients with mantle cell lymphoma who are failed or relapsed after remission or intolerated to Bruton's tyrosine kinase (BTK) inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Per 2017 revised WHO lymphoma classification criteria, subject must have diagnosed with MCL.
2. At least one measurable lesion.
3. Subjects who have previously received the treatment regimen containing anti-CD20 and at least one BTKi treatment failed or relapsed after remission or intolerated; Or Subjects who have previously received BTK inhibitors treatment failed or relapsed after remission or intolerated, and are not suitable for treatment with anti-CD20.
4. ECOG≤2.
5. Adequate hematologic function.
6. Adequate hepatic and renal function.
7. Willingness of men and women of reproductive potential (defined as following menarche and not postmenopausal [and 2 years of non-therapy-induced amenorrhea] or surgically sterile) to observe conventional and effective birth control.

Exclusion Criteria:

1. Received non-covalent BTK inhibitor treatment.
2. Subjects who have received the following treatments within 4 weeks or 5 half-lives before the first dose of Rocbrutinib: Antitumor therapies including myelosuppressive chemotherapy, targeted therapy, biological therapy and/or immunotherapy; Any investigational treatment; Patients who have undergone major surgery, severe trauma or radiotherapy.
3. Subjects who have received the following treatments within 2 weeks before the first dose of Rocbrutinib: Steroids or traditional herbal medicine for antitumor purposes; Strong and moderate CYP3A inhibitors and inducers; All drugs that may cause QTc interval prolongation or torsional tachycardia.
4. Disease states where clinical manifestations may be difficult to control, including HIV, HBV, HCV, syphilis positive or active bacterial and fungal infections.
5. Disease affects the central nervous system.
6. Any gastrointestinal conditions that may severely affect the study drug absorption or pharmacokinetic parameters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | Up to 24 Months
  To assess the anti-tumor activity of Rocbrutinib based on overall response rate (ORR) as assessed by Independent Reading Committee (IRC).

SECONDARY OUTCOMES:
Overall Response Rate | Up to 24 Months
  To assess the anti-tumor activity of Rocbrutinib based on overall response rate (ORR) as assessed by investigator.
Complete remission rate | Up to 24 Months
  To assess the preliminary anti-tumor activity of Rocbrutinib based on complete remission rate (CR) as assessed by investigator and IRC.
Progression Free Survival | Measured from the date of first dose of study drug to the date of earliest disease progression or death or last visit, and assessed up to 24 months.
  To assess the preliminary anti-tumor activity of Rocbrutinib based on Progression Free Survival (PFS) as assessed by investigator and IRC.
Overall survival | Measured from the date of date of first dose to the date of death or last visit, and for up to 5 years after the last subject is enrolled.
  To assess the preliminary anti-tumor activity of Rocbrutinib based on Overall survival (OS) as assessed by investigator and IRC.
Duration of Response (DOR) | Measured from the date of the first remission to the date of earliest disease progression or death, and assessed up to 24 months.
  To assess the preliminary anti-tumor activity of Rocbrutinib based on Duration of response (DOR) as assessed by the Investigator and IRC.
Time to Response (TTR) | Measured from the date of the first dose of study drug to the date of earliest response, and assessed up to 6 months.
  To assess the preliminary anti-tumor activity of Rocbrutinib based on Time to response (TTR) as assessed by the Investigator and IRC.
Safety Assessment | From first dose of study drug to 28 days after last dose of study drug
  To evaluate the safety of Rocbrutinib by assessing incidence and severity of treatment-emergent adverse events as determined by CTCAE v5.0
Maximum Observed Plasma Concentration (Cmax) | Up to 24 hours post dose
  Pharmacokinetics (PK) As Assessed By Maximum Observed Plasma Concentration (Cmax) Of Rocbrutinib
Area Under The Plasma Concentration Time Curve From Time 0 To The Time Of The Last Quantifiable Concentration (AUC0-t) | Up to 24 hours post dose
  PK As Assessed By Area Under The Plasma Concentration Time Curve From Time 0 To The Time Of The Last Quantifiable Concentration (AUC0-t) of Rocbrutinib
Maximum Observed Plasma Concentration (Tmax) | Up to 24 hours post dose
  PK As Assessed By Time To Maximum Observed Plasma Concentration (Tmax) Of Rocbrutinib
Half-life period (T1/2) | Up to 24 hours post dose
  PK As Assessed By Time To Half-life period (T1/2) Of Rocbrutinib
Quality of life (QoL) | Up to 24 Months
  Quality of life Assessed By the European Organization for Research and Treatment of Cancer core quality of life (EORTC QLQ-C30) questionnaire (The total score ranges from 30 to126, Items 29 and 30 are scored from 1 to 7 points, and other items are scored from 1 to 4 points. Except for items 29 and 30, the higher value, the worse QoL.)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, MD, PhD, Study Chair — Peking University Cancer Hospital & Institute
Locations (43):
- China (43):
  - Anhui provincial cancer hospital, Hefei, Anhui
  - The first affiliated hospital of Anhui medical university, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The first affiliated hospital of Chongqing mediacal university, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fujian Medical university union hospital, Fuzhou, Fujian
  - The first affiliated hospital of Xiamen university, Xiamen, Fujian
  - Gansu provincial cancer hospital, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Meizhou people'shospital, Meizhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The fourth hospital of Hebei medical university, Shijiazhuang, Hebei
  - Harbin First Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan provincial people's hospital, Zhengzhou, Henan
  - The first affiliated hospital of Zhengzhou university, Zhengzhou, Henan
  - Hunan cancer hospital, Changsha, Hunan
  - Jiangsu cancer hospital, Nanjing, Jiangsu
  - Jiangsu province hospital, Nanjing, Jiangsu
  - The first affiliated hospital of Nanchang university, Nanchang, Jiangxi
  - The second hospital of dalian medical university, Dalian, Liaoning
  - Shengjing hospital of China medical university, Shenyang, Liaoning
  - The first hospital of China medical university, Shenyang, Liaoning
  - Qilu hospital of Shandong university, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - West China School of Medicine, Chengdu, Sichuan
  - Tianjin Hematonosis Hospital, Tianjin, Tianjin Municipality
  - Tianjin medical university cancer hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Affiliated hospital of hebei university, Baoding
  - Beijing Boren Hospital, Beijing
  - Beijing Friendship hospital, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - Sichuan Cancer Hospital, Chengdu
  - The First People's Hospital of Foshan, Foshan
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Sun Yat-sen Memorial Hospital, Guangzhou
  - The First Affiliated Hospital of Soochow University, Suzhou
  - The first affiliated hospital of Wenzhou medical university, Wenzhou
  - Hubei Cancer Hospital, Wuhan
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: No